CLINICAL TRIAL: NCT00418990
Title: Effect of a Randomized Trial of Multivitamin-Mineral Supplementation on Standardized Assessment of Academic Performance in Elementary School Children
Brief Title: Effect of Vitamins on Academic Performance of School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Rutgers University (Other)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-681
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Last update posted 2007-01-05 (Estimated); Status verified 2007-01

CONDITIONS: Malnutrition
Keywords: Multivitamin; Academic performance
MeSH Terms: conditions — Malnutrition | interventions — Geritol

INTERVENTIONS:
Drug: Multivitamin/Mineral supplements

SUMMARY:
The purpose of this clinical trial is to determine if administration of a daily chewable multivitamin-mineral supplement (Monday - Friday when school is in session) given to children (third through sixth graders) during the academic school year will lead to improved academic performance.

DETAILED DESCRIPTION:
SUMMARY OF PROPOSED PROJECT IN LAY TERMS:

The purpose of this clinical trial is to determine if administration of a daily chewable multivitamin-mineral supplement (Monday - Friday when school is in session) given to children (third through sixth graders) during the academic school year will lead to improved academic performance.

Letters will be mailed to parents of all entering third through sixth graders in the Newark School System in August, explaining the study and containing a self-addressed stamped postcard. The postcard will allow parents to express whether or not they wish to be invited to an informational meeting. Location of the meeting will be determined in consultation with the school system. During the meetings, dinner will be served and further information about the study will be disseminated. At the end of the meetings, the informed consent/assent process will be undertaken by the PI and study personnel. Children who are currently taking multivitamins at least five days per week or did not take the Assessment of Skills and Knowledge exam at the completion of the third (3rd) grade will be excluded. Children taking a multivitamin less than five days per week will be eligible if they discontinue its use during the study period. Presentations at the Parent/Teacher Conferences at the beginning of the academic year by Investigators will also be utilized to help answer questions about participation and identify potential volunteers.

Once informed consent and assent have been received, all children will be randomly assigned to receive either 2 tablets of a multivitamin-mineral supplement or 2 tablets of an inactive placebo daily (Monday - Friday when school is in session) in school. The multivitamin-mineral supplement will be analyzed by the United States Pharmacopeial Convention, Inc. (USP) to assure the supplement (1) contains the declared vitamin and mineral ingredients on the product label, (2) contains the amount or strength of ingredients declared on the product label, (3) meets requirements for limits on known contaminants, and (4) otherwise conforms to the USP monograph for the article (Appendix F). Children will receive these tablets in ID numbered envelopes distributed by teachers or study personnel with the morning snacks during the school week for a seven (7) to eight (8) month period in the school year. Pill counts and attendance records will help assess treatment compliance. Participants will receive $10 and free vitamins for one year following the completion of the study.

In order to assess academic performance, information on grade point average, missed days of school and performance on the State of New Jersey's standardized Assessment of Skills and Knowledge (ASK) exam for grades 3, 4, 5 and 6 for each participating child will be obtained from the student record. Demographic information including height, weight, body mass index, age, race and gender will be collected on all children. Height and weight will be measured in the schools by study personnel at the beginning and end of the study period. On a subset of children (n=250, the Block Food Frequency Questionnaire for children will be administered by study personnel at the beginning of the study period to ascertain a record of nutritional intake.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in third through sixth grades in the Archdiocese of Newark School System during 2004-2005 academic year.
* Completion of the Assessment of Skills and Knowledge Exam in 2003

Exclusion Criteria:

* Known allergy to any ingredients of the multivitamin.
* Currently taking a multivitamin on a regular basis.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1600
Dates: Start 2003-08; Study Completion 2005-11

PRIMARY OUTCOMES:
Assessment of Skills and Knowledge Exam

SECONDARY OUTCOMES:
Gradepoint average
Absenteeism
Incidents of misbehavior

CONTACTS AND LOCATIONS:
Overall Officials: Adam ' Perlman, MD, MPH, Principal Investigator — University of Medicine & Dentistry of New Jersey
Locations (1):
- University of Medicine & Dentistry of New Jersey, Newark, New Jersey, United States